CLINICAL TRIAL: NCT06316583
Title: Clinical Study of Dry Needling on Myofascial Trigger Points Treatment for Primary Dysmenorrhea and Preliminary Investigation of Its Relevance to Acupoints
Brief Title: Clinical Study on Dry Needling for Primary Dysmenorrhea and Its Preliminary Correlation With Acupoints
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Collaborators: Beijing Municipal Health Commission (Other Government)
Responsible Party: Principal Investigator, Yanxia Sun, Principal Investigator, Beijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BJH-001
Record Dates: First submitted 2024-03-05; First posted 2024-03-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-03

CONDITIONS: Trigger Point Pain, Myofascial; Acupuncture; Primary Dysmenorrhea
Keywords: trigger points, dry-needling, primary dysmenorrhea
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Acupuncture Therapy

STUDY DESIGN:
Intervention Model Description: Using a single-center randomized controlled patient-blind study design, 150 eligible participants are randomly assigned to three groups: a placebo group (sham trigger point needling), a dry-needling trigger points treatment (TrP-DN)group, and a traditional acupuncture group. Compared to the placebo group, this study assesses the effects of TrP-DN and traditional acupuncture on pain and quality of life for primary dysmenorrhea patients, as well as their long-term outcomes. Additionally, the study observes their impact on inflammatory factors and local uterine blood flow, aiming to explore the mechanisms underlying TrP-DN and traditional acupuncture treatments for PD.
Who Masked: Participant, Outcomes Assessor
Masking Description: This experiment is a single-blind study where randomization occurs centrally through an online data management system after collecting baseline data from participants. A designated research coordinator manages the randomization process and facilitates communication among research personnel. Due to the nature of the intervention, operators are aware of the group assignments, but evaluators, unaware of these assignments, assess and collect baseline, post-treatment, and follow-up data. Since none of the participants have received any prior acupuncture or trigger point dry needling treatments, using a scalable sham needle on the same trigger points ensures blinding by simulating the effects of actual treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- dry-needling trigger points treatment (TrP-DN) (Experimental): Firstly, use pressure techniques to diagnose trigger points on the rectus abdominis and oblique muscles, which typically present as distinct tender points and palpable muscle tension bands. Deep pressure on these points may induce referred pain. Procedure: Begin by disinfecting the treatment sites. Use a traditional acupuncture needle (0.35×50mm) to repeatedly stimulate the designated point until muscle soreness and localized twitching are felt. If participants experience lower back pain, trigger points on the back can also be targeted, located bilaterally from the twelfth thoracic vertebra to the third lumbar vertebra
  Interventions: Other: TrP-DN and Acupuncture
- acupuncture group (Experimental): Acupuncturists use acupuncture point needling for treating PD, focusing primarily on key acupoints from the Foot Taiyin Spleen Meridian, Conception Vessel, Foot Taiyang Bladder Meridian, Foot Yangming Stomach Meridian, and Foot Shaoyin Kidney Meridian. Commonly selected points include Taichong, Xuehai, Zusanli, Yanglingquan, Guanyuan, Uterus, and Sanyinjiao. After routine disinfection, a #32 fine needle is quickly inserted and retained for 30 minutes per session
  Interventions: Other: TrP-DN and Acupuncture
- placebo control group (Sham Comparator): Subjects undergo the same diagnostic and therapeutic procedures as the TrP-DN group but using a 'sham' needling technique. The sham needling is administered by the same expert as the real needling, with retention time and treatment frequency matching those of the genuine needling group. A retractable sham needle apparatus is used without piercing the skin.
  Interventions: Other: TrP-DN and Acupuncture

INTERVENTIONS:
Other: TrP-DN and Acupuncture — Treatment is conducted by pain specialists and acupuncturists, each having over 5 years of relevant work experience. The treatment occurs within the three weeks leading up to menstruation, administered once a week for a total of three sessions. Additionally, participants are to engage in abdominal stretching exercises starting from the treatment day. These exercises are to be done 3-5 times daily, with each session lasting approximately 2 minutes, and this regimen is to continue for one month. If participants experience significant pain during menstruation, they may take NSAIDs orally for symptomatic relief.

SUMMARY:
Primary dysmenorrhea refers to menstrual pain not caused by pelvic organic lesions, commonly seen in young women, significantly affecting patients' quality of life. Dry needling therapy targeting myofascial trigger points for primary dysmenorrhea has been preliminarily applied in clinical settings. However, related research is limited with questionable quality, hindering its widespread clinical application. Furthermore, is there a connection between myofascial trigger points in dry needling and acupuncture acupoints in terms of selection and mechanism of action? Could this be a new interpretation of acupuncture theory? These are important questions that have garnered widespread attention. This study employs a randomized patient-blinded controlled design, enrolling primary dysmenorrhea patients aged 18 to 30 years. They are randomly divided into three groups: the trigger point dry needling group, traditional acupuncture treatment group, and trigger point sham needle (placebo) group. Changes in pain levels, quality of life scores, inflammatory factor levels, and local blood flow before and after treatment among the three groups are observed. The aim is to assess the therapeutic effects of dry needling trigger points and acupuncture treatments on primary dysmenorrhea and explore their potential mechanisms of action. By comparing the differences and similarities between dry needling trigger points and acupuncture treatments in terms of acupoint selection, treatment effects, and potential mechanisms of action, this study seeks to preliminarily explore the feasibility of integrating trigger point theory into the meridian 'acupoint' theory, laying the foundation for a modern interpretation of acupuncture

DETAILED DESCRIPTION:
Using a single-center, randomized, single-blind study design, 150 eligible subjects were randomly divided into three groups: placebo group (pseudo-acupuncture trigger point group), TrP-DN treatment group, and traditional acupuncture treatment group. Compared with the placebo control group (trigger point sham needle group), the study evaluated the effects of TrP-DN and traditional acupuncture treatment on pain, quality of life, and long-term prognosis of PD patients. The study also observed their effects on inflammatory factors and local uterine blood flow, exploring the possible mechanisms of TrP-DN and traditional acupuncture treatment for PD.

Further observations were made on the differences and similarities between conventional TrP-DN and traditional acupuncture treatment in terms of point selection, treatment effects, and their effects on inflammatory factors and local uterine circulation. The study aimed to explore the relationship between the trigger point theory and the theory of meridians and acupoints, providing a research basis for integrating TrP-DN into traditional acupuncture theory.

ELIGIBILITY:
Inclusion Criteria:

1. All participants diagnosed explicitly by a gynecologist as having primary dysmenorrhea without pelvic organic lesions.
2. Aged between 18 and 30 years.
3. A history of cyclical menstrual pain for more than 2 years.
4. Pain greater than 30mm on the Visual Analog Scale (VAS, 0-100mm).
5. Participants must sign an informed consent form and be willing to undergo acupuncture treatment and cooperate to complete the relevant procedures of this trial.

Exclusion Criteria:

1. Those suffering from secondary dysmenorrhea or any other reproductive and urinary system diseases, such as endometriosis.
2. A history of pregnancy, miscarriage, or planning for pregnancy. Individuals with skin infections on the abdomen and lower back.
3. Past use of acupuncture therapy or other needling treatments.
4. Those with a history of mental illness and severe diseases of the heart, liver, brain, kidneys, hematopoietic system, etc.
5. Within the past 6 months, individuals referred to pain clinics, those who have used pain relievers like morphine or pethidine, or those allergic to NSAIDs. Also, those currently taking or receiving anticoagulant medications.
6. Individuals who have had adverse reactions to acupuncture (e.g., fainting).

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
mean intensity of pain | menstrual cycle before treatment, the month after treatment, the second month after treatment,
  Participants are asked to mark their intensity of pain using Visual Analog Scale during period time a 100mm horizontal line, with the ends of the line representing the extreme expressions of pain (no pain to maximum pain).The mean intensity of all days with menstrual pain is used for the analysis

SECONDARY OUTCOMES:
mean intensity of painscale during period a 100mm horizontal line, with the ends of the line representing the extreme expressions of pain (no pain to maximum pain).The mean intensity of all days with menstrual pain is used for the analysis | menstrual cycle one year after treatment
  Participants are asked to mark their intensity of pain on Visual Analog Scale (0 no pain and 100mm refer to worst pain)
Short Form Health Survey | menstrual cycle before treatment, the month after treatment, the second month after treatment, and one year after treatment
  Short Form Health Survey-36 (The minimum score for each question is 0, indicating the worst possible health status or quality of life,The maximum score for each question is 100, indicating the best possible health status or quality of life.)
Global Rating of Change Scale | menstrual cycle at the month after treatment, the second month after treatment, and one year after treatment
  Global Rating of Change Scale(GROC)[It typically ranges from -5 to +5, with 0 representing no change, -5 indicating a very marked worsening, and +5 indicating a very marked improvement]
the amount of NSAIDs used | menstrual cycle before treatment, the month after treatment, the second month after treatment, and one year after treatment
  the total amount of NSAIDs used during period
the frenquecy of NSAIDs used | menstrual cycle before treatment, the month after treatment, the second month after treatment, and one year after treatment
  the total times of NSAIDs used during period
inflammatory factors | menstrual cycle before treatment, the same month after treatment, and during the second month after treatment (specifically on the second day of the menstrual cycle as recommended in the study)
  the study uses ELISA to measure specific inflammatory markers in participants at different time points related to their menstrual cycles before and after treatmen.The inflammatory factors examined are based on previous research results and include prostaglandin F2-α (PGF2-α), C-reactive protein (CRP), interleukin-6 (IL-6), and interleukin-8 (IL-8).
local uterine blood flow：Doppler Systolic/Diastolic (S/D) Ratio | the same day of the menstrual cycle (specifically recommended on the second day of the menstrual cycle) before treatment, during the same month after treatment, and during the second month after treatment.
  Using transabdominal color Doppler ultrasound to measure the blood flow of the uterine artery at the lateral border of the cervix: The S/D ratio provides information about the ratio of systolic (peak) to diastolic (minimum) velocities in the blood vessel. A higher S/D ratio indicates higher vascular resistance, while a lower ratio suggests lower resistance.
local uterine blood flow：Pulsatility Index (PI) | the same day of the menstrual cycle (specifically recommended on the second day of the menstrual cycle) before treatment, during the same month after treatment, and during the second month after treatment.
  Using transabdominal color Doppler ultrasound to measure the blood flow of the uterine artery at the lateral border of the cervix:The PI provides information about the vascular resistance. A higher PI indicates higher resistance to blood flow, which can be seen in conditions such as vasoconstriction or occlusion. Conversely, a lower PI suggests lower resistance, which can be seen in conditions such as vasodilation or increased blood flow.
local uterine blood flow：The Resistance Index (RI) | the same day of the menstrual cycle (specifically recommended on the second day of the menstrual cycle) before treatment, during the same month after treatment, and during the second month after treatment.
  The Resistance Index (RI) is a parameter used in Doppler ultrasound to assess vascular resistance. It is calculated as the difference between the peak systolic velocity (PSV) and the end diastolic velocity (EDV), divided by the peak systolic velocity. The RI provides information about vascular resistance. A higher RI indicates higher vascular resistance, which may occur in conditions such as vasoconstriction or occlusion. Conversely, a lower RI suggests lower resistance, which may occur in conditions such as vasodilation or increased blood flow.
Number of Participants with adverse effects with treatment | through study completion, an average of 2 year
  This includes unexpected reactions or uncomfortable symptoms, with a particular focus on complications related to acupuncture. All adverse events reported by participants will be documented in the Case Report Form (CRF).

OTHER OUTCOMES:
Assessing Participants Expectations of Outcomes of Complementary and Alternative Medicine Treatments | before treatment
  The Acupuncture Expectancy Scale (The scores for each item can be adjusted based on the individual being assessed, and the final score can reflect the individual's overall expectancy and confidence levels regarding acupuncture treatment.)
Rate of same points used between dry-needling group and traditional acupuncture group | through study completion, an average of 2 year
  The same acupuncturist compare the trigger points of the TrP-DN group with the sham needle group to determine if they are indeed acupuncture points, and specify their exact names. Record the acupuncture points used for the participants in the needling group and indicate them

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhen, Study Chair — Beijing Hospital; Yanxia Sun, Principal Investigator — Beijing Hospital
Locations (1):
- Yanxia Sun, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
All data relevant to the study will be included in a published article or uploaded as supplemental information. Our protocol is available on Clinicaltrial.gov and all search strategies will be available in supplemental materials.

REFERENCES:
- [Derived] Sun Y, Yang L, Zhu L, Zhang S, Cheng W, Lin L, Li W, Li M, Zhao X, Guo J, Hua Z. Efficacy of Myofascial Trigger Point Dry Needling in Treatment of Primary Dysmenorrhea: A Study Protocol for a Three-Arm Randomized Controlled Trial. J Pain Res. 2025 Sep 5;18:4623-4633. doi: 10.2147/JPR.S537971. eCollection 2025. PMID 40933501